CLINICAL TRIAL: NCT06314022
Title: Design of a Mobile Application to Improve the Quality of Colonoscopy and Its Implementation in Colorectal Cancer Screening Program: a Randomized Multicenter Study (PrepColon APP Study)
Brief Title: A Mobile Application to Improve the Quality of Colonoscopy in Colorectal Cancer Screening Program (PrepColon APP)
Acronym: PREPCOLON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Mª Henar Núñez Rodriguez, MD PhD, Principal Investigator, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-PI113
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Premalignant Colon Lesions
Keywords: quality colonoscopy; colorrectal cancer screening; mobile application
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized into two groups according to the instructions given to perform the preparation of the colon prior to colonoscopy: group A: perform the preparation with the written instructions delivered in the consultation and group B: they will be given the instructions in writing and will also be indicated how to install the APP.
Who Masked: Investigator
Masking Description: Patients who agree to participate in the study are randomized by a 1:1 block computer program (an attempt will be made to balance the groups according to the type of laxative) into two groups: group A: control group, which receives the standard information given in writing, and group B: APP group, which receives the standard information together with the mobile application individually adapted to the scheduled colonoscopy appointment and the type of laxative.
  Patients scheduled for a screening colonoscopy will be contacted by telephone, those who agree to participate will be scheduled with the nurse, after giving their consent they are randomized. Group B will indicate how to download the APP and its management. The endoscopist performing the examination is blind for randomization and will assess colon cleansing according to the Boston Bowel Scale (Lai EJ. et al Gastroinest Endosc 2009).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): which receives the standard information given in writing,
- APP group (Experimental): Group which receives the standard information together with the mobile application individually adapted to the scheduled colonoscopy appointment and the type of laxative.
  Interventions: Other: Mobile application for colonoscopy preparation instructions

INTERVENTIONS:
Other: Mobile application for colonoscopy preparation instructions — The APP will also consider the comorbidities and drugs of each patient. It can be adapted to the different types of laxative (4, 2 or 1 litre) and notify the need to discontinue anticoagulant and/or antiplatelet treatments by contacting with the primary care physician. Additionally, the application may ask short questions to the patient to control the laxative intake instruction. The user must confirm the appointment 48 hours in advance.
  Arms: APP group

SUMMARY:
Colonoscopy is the gold standard for the diagnosis and resection of preneoplastic lesions, allowing the prevention of colon cancer. A colonoscopy is more efficient with proper preparation of the colon, as it allows for a higher rate of adenoma detection and cecal intubation. In routine practice, up to 30% of colonoscopies are poorly prepared and 11% of patients do not show up for their appointment. Adenomas not visualized in the initial colonoscopy due to poor preparation reached 68% and the rate of undetected cancers was 66.7%. A proper colon cleanse is conditioned by different factors; among them, failure to comply with the diet and take laxatives poses 5 times the risk of having a deficient colon preparation. The purpose of our study is the design and implementation of an app that facilitates the preparation of colonoscopy and evaluates its impact on compliance with diet and laxative intake.

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODS

Study Design:

Phase 1: Design of the mobile application (APP): The APP will be designed in a participatory manner by the research team of the project, formed by doctors, nurses, statisticians and telecommunications engineers. The application should be usable with both Android and iOS devices, so we will use the Flutter framework to build apps for different platforms with a single code base.

When arranging a colonoscopy, the patient will install the APP on their mobile phone and indicate the date and time of the test. The APP will be responsible for supporting the preparation of the colon cleansing, for which, in addition to being able to visualize the corresponding information, it will make use of notifications to show diet reminders and laxative intakes.

More specifically, these could be some notifications:

* (3 days before the appointment) - Notification of start of preparation with a low fibre diet
* (24 hours before the appointment) - Notification of .laxative intake..

The APP will also consider the comorbidities and drugs of each participant. It can be adapted to the different types of laxative (4, 2 or 1 litre) and notify the need to discontinue anticoagulant and/or antiplatelet treatments by contacting with the primary care physician. Additionally, the application may ask short questions to control the laxative intake instruction. The user must confirm the appointment 48 hours in advance. The design of the APP aims to be intuitive and easy to use by the target population (50-69 years), allowing to adapt the font size and zoom in on the images to facilitate the visualization of the information.

The APP will be multilingual for English and Spanish, and others may be incorporated if deemed necessary. An agile and iterative methodology of software development will be followed as SCRUM in the realization of the APP. Thus, sprints of about 3 weeks will be planned with delivery of functional software that will progressively incorporate the different functionalities planned for the APP.

Phase 2: Re-evaluation of the APP after the inclusion of 30 patients, the APP will be re-evaluated through a usability questionnaire and adjustments and changes will be made if necessary

Phase 3: Prospective, multicentre and randomized study in asymptomatic patients between 50 and 69 years who attend screening colonoscopy after a positive FIT >100 ng / ml)

The study will be carried out in the Digestive Service of 3 hospitals in Castilla y León: Virgen de la Concha Hospital in Zamora, Medina del Campo Hospital and Río Hortega University Hospital in Valladolid. Participants will be randomized into two groups according to the instructions given to perform the preparation of the colon prior to colonoscopy: group A: perform the preparation with the written instructions delivered in the consultation and group B: the investigators will give the instructions in writing and will also indicate how to install the APP to the participants.

ELIGIBILITY:
Inclusion Criteria:

* -Subjects between 50-69 years old from the CRC screening program with FIT (>100ng/ml).
* Informed consent granted in writing

Exclusion Criteria:

* Refusal to give informed consent.
* Those who do not have a smartphone with a minimum version of the operating system (Android 4.4 or iOS 14, which cover more than 99% of the terminals in use)
* Symptomatic patients
* Subjects at elevated risk of CRC due to family history or inherited polyposis diseases or inflammatory bowel disease

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Compliance with the diet and intake of laxatives with the use of a mobile application | at the moment of the procedure
  Questionnaire about ASSESSMENT OF DIET COMPLIANCE (number of portions 0->2, higher points means worse outcome):
  Have you followed the diet without fiber the 3 days prior to preparation: YES/ NO
  * Have you eaten fruits, vegetables and legumes? number of portions 0 1 2 >2
  * Have you eaten whole grain products? number of portions 0 1 2 >2
  * Have you eaten meats and sausages? number of portions 0 1 2 >2
  * Have you eaten blue fish? number of portions 0 1 2 >2
  * Have you eaten nuts? number of portions 0 1 2 >2
  * Have you eaten anything solid in the last 24 hours? yes/ no
Evaluate the quality of colon cleansing with mobile application as an experimental factor | at the moment of the procedure
  The endoscopy will assess colon cleansing according to the Boston Bowel Scale (BBPS) uses a 4-point rating system (0-3) applied to each of the 3 segments of the colon (right, transverse, left) to assess colon cleanliness during the withdrawal phase of colonoscopy, after all cleaning maneuvers have been performed. (0 worse outcome and 3 best outcome)
Assessment of the usability of the APP | at the moment of the procedure
  A questionare: System Usability scale (SUS), ten question about usability with Five responses ranging from Strongly Agree to Strongly Disagree
Compliance with the laxative intake with the use of the mobile application | At the moment of the procedure
  Questionnaire to EVALUATE COMPLIANCE WITH TAKING THE LAXATIVE: questions like at • --Type of laxative: (name):
  * Colonoscopy appointment (time) Morning / Afternoon
  * Start of taking the laxative: time:
  * End of taking the laxative (How many hours ago did you finish taking the laxative before the appointment?
  * Have you taken all of the laxative?
  * How much liquid have you drunk?
  * How many shots have you done it in? How much liquid does each drink?

SECONDARY OUTCOMES:
Assessment of the difficulty of the preparation instructions | at the moment of the procedure
  quesionnaire: EVALUATION OF THE COMPRESSION OF THE INSTRUCTIONS GIVEN: scale from 0 to 10 (0:worse outcomes and 10: best outcomes)
Evaluate colonoscopy quality indicators: | at the moment of the procedure and after one month with the histological results
  Adenoma detection rate (ADR) is the percentage of patients with at least one histologically proven adenoma or carcinoma
Evaluate attendance at the scheduled colonoscopy appointment | at the moment of the colonoscopy
  Attendance or not to colonoscopy appointment
Evaluate colonoscopy quality indicators | at the moment of the colonoscopy
  Cecal intubation rate is the percentage of patients with completed colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Henar Nuñez Rodriguez, MDPhD, Principal Investigator — Hospital Universitario Rio Hortega
Locations (1):
- Hospital Universitario Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No